CLINICAL TRIAL: NCT02992873
Title: The Scandinavian AED and Mobile Bystander Activation Trial - a Randomized Controlled Trial
Brief Title: The Scandinavian AED and Mobile Bystander Activation Trial
Acronym: SAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Hollenberg, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT2
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Cardiac Arrest, Sudden
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Layperson allocated to fetch an AED and start CPR (Experimental): In the intervention group mobile lifesavers will be directed to fetch the nearest AED and then attach it to the victim of OHCA. At least 1 volunteer will be directed to start CPR only
  Interventions: Device: Layperson allocated to start CPR and fetch nearest AED
- Layperson allocated to start CPR (Active Comparator): In the control group all mobile lifesavers will be directed to the patient to start CPR.
  Interventions: Device: Layperson allocated to start CPR

INTERVENTIONS:
Device: Layperson allocated to start CPR and fetch nearest AED — Dispatching laypersons to fetch an AED and start CPR in out-of-hospital cardiac arrest
  Other Names: Dispatch to start CPR and fetch nearest AED
  Arms: Layperson allocated to fetch an AED and start CPR
Device: Layperson allocated to start CPR — Dispatching laypersons to start CPR out-of-hospital cardiac arrest
  Other Names: Dispatch to start CPR
  Arms: Layperson allocated to start CPR

SUMMARY:
Sudden cardiac death is a major health problem in the western world. In Europe alone nearly 300 000 patients are affected annually. The majority of victims suffering from an Out-of-Hospital Cardiac Arrest (OHCA have an initial cardiac rhythm that can be treated by means of defibrillation. In most emergency medical systems (EMS) time to defibrillation is too long and survival averages 10 %.However, when laymen operated Automated External Defibrillators (AEDs) are used within the first minutes, 7 out of 10 may survive.

The aim of "The Scandinavian AED and Mobile Bystander Activation" (SAMBA) trial is to evaluate if a Mobile Phone Positioning system and a smartphone application will increase the proportions of patients with an attached Automated External Defibrillator (AED) before arrival of the Emergence Medical System (EMS). Mobile phone technology and a smartphone application will be used identify and recruit nearby CPR-trained lay people and automated external defibrillators (AEDs) to patients suffering out-of-hospital cardiac arrest (OHCA). The system is currently running in Stockholm Sweden and in the Gothenburg region.

DETAILED DESCRIPTION:
Early defibrillation in out-of-hospital cardiac arrest is associated with high survival rates. If the operator at the dispatch center suspects an out-of-hospital cardiac arrest he or she will activate the mobile positioning system (MPS) wich is integrated in the operators computer environment.

After activation, the system will locate all CPR-trained volunteers nearby the suspected OHCA. By computer based 1:1 randomization lay volunteers will be alerted and dispatched in 50 % of all suspected OHCAs in where the system is triggered by the dispatchers. In the intervention group, the activation of the system is supposed to result in lay volunteers to be alerted and directed to fetch the nearest AED and commence early defibrillation. Dependent on geographical and logistical circumstances, at a minimum one lay volunteer or more will be alerted to provide bystander CPR only.

In the control group the MPS will be activated and lay responders will be dispatched to suspected OHCA to perform CPR only. In both groups the ordinary EMS services are dispatched in a regular fashion.

ELIGIBILITY:
Inclusion Criteria:

* All EMS-treated OHCAs within the Stockholm County, Copenhagen and VGR area and in whom the mobile positioning system is activated at the emergency dispatch center

Exclusion Criteria:

* Crew witnessed OHCAs
* Patients <8 years of age
* OHCAs due to trauma, intoxication, or suicide
* OHCAs not treated by the EMS due to ethical reasons or obvious signs of death.
* No OHCA cases

Ages: 8 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 815 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with AED attached prior to arrival of EMS, fire or police services. | 12 months
  Attached public AED before arrival of EMS or first responders (fire, police).

SECONDARY OUTCOMES:
Proportion of patients with bystander CPR prior to arrival of EMS, fire or police services. | 12 months
  Any bystander CPR before arrival of EMS, fire or police services
Proportion of patients defibrillated before arrival of EMS, fire or police services arrival. | 12 months
  Use of (defibrillation) AED before EMS (ambulance fire and police) arrival.

OTHER OUTCOMES:
Adverse events prehospital | 12 months
  All adverse events reported at a prehospital stage will be collected and presented as minor or major events related to lay persons participating as mobile phone dispatched rescuers events related to patients. Minor events are negative safety events with the potential to harm the lay rescuer or patient such as technical malfunction or dispatcher related communication failure. Major events are negative events that actually harms the lay rescuer or OHCA patient due to system malfunction, such as unsafe scene or violation of integrity.
Proportion of CRP by mobile phone dispatched lay volunteers. Both study groups combined. | up to 12 months
  Additional (total) effect of mobile phone dispatched lay volunteers in both study groups (observational)
Adverse advents in relation to SMS -alerts, AED use and lay responders | 12 months
  Adverse events concerning the dispatch of lay volunteers
Proportion of AED attachment prior to the EMS by mobile phone dispatched lay volunteers. Both study groups combined. | 12 months
  Additional (total) effect of mobile phone dispatched lay volunteers in both study groups (observational)

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ringh, MD, PhD, Principal Investigator — Karolinska Institutet; Jacob Hollenberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Västra Götaland, Gothenburg
  - Stockholm, Sweden, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berglund E, Hollenberg J, Jonsson M, Svensson L, Claesson A, Nord A, Nordberg P, Forsberg S, Rosenqvist M, Lundgren P, Hogstedt A, Riva G, Ringh M. Effect of Smartphone Dispatch of Volunteer Responders on Automated External Defibrillators and Out-of-Hospital Cardiac Arrests: The SAMBA Randomized Clinical Trial. JAMA Cardiol. 2023 Jan 1;8(1):81-88. doi: 10.1001/jamacardio.2022.4362. PMID 36449309